CLINICAL TRIAL: NCT00408915
Title: Double-blind, Placebo-controlled, Randomized, Multicentre Phase II/III Study to Evaluate the Efficacy and Safety of Lisuride, Applied Subcutaneously by Means of a Minipump in Patients With Advanced Parkinson's Disease Refractory to Conventional Oral Therapy
Brief Title: Continuous Application of Lisuride in Parkinson's Disease by Subcutaneous Infusion
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Axxonis Pharma AG (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CALIPSO; EudraCT number:; 2005-001006-12
Record Dates: First submitted 2006-12-05; First posted 2006-12-07 (Estimated); Last update posted 2012-03-07 (Estimated); Status verified 2012-03

CONDITIONS: Parkinson's Disease
Keywords: Lisuride; Continuous Dopaminergic Stimulation; Motor Fluctuations; Off-Times; Troublesome Dyskinesia; Parkinson's Disease with motor fluctuations with OFF periods and/or troublesome dyskinesias of more than four hours per day
MeSH Terms: conditions — Parkinson Disease

INTERVENTIONS:
Drug: Continuous Subcutaneous Lisuride Infusion

SUMMARY:
The aim of the study is to evaluate the long-term efficacy, local tolerability and safety of Lisuride applied as subcutaneous infusion compared to placebo in patients with advanced Parkinson's disease with motor fluctuations and "OFF" periods refractory to conventional treatment.

DETAILED DESCRIPTION:
The current CALIPSO study investigates the efficacy of a continuous lisuride infusion against the optimized previous oral therapy in patients experiencing motor fluctuations with OFF periods and/or strenuous dyskinesias of more than four hours per day.

The controlled core study is scheduled to last six weeks. Within the study the previous oral therapy will either be continued in a capsule/blinded design (while a placebo infusion is going on concurrently) or the oral therapy is substituted by lisuride infusion (while placebo capsules are administered at the same time).

After the controlled core study all patients whose condition has not worsened during the study (meaning those patients of the placebo infusion group as well, who were treated during the core study just as they were before), will be given the chance to continue with the infusion therapy with lisuride in an open extension phase.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's disease for at least 3 years (diagnosis based on the UK Brain Bank Criteria)
* Presence of motor fluctuations (wearing-off or other "OFF" periods) and / or presence of troublesome dyskinesia, with a total daily minimum of at least 4 hours, despite optimized oral anti-parkinsonian therapy
* Stable levodopa intake, i.e. at least four doses of levodopa per day
* Stable dosing of all other anti-parkinsonian drugs, such as dopamine agonists, COMT- and MAO-B inhibitors, amantadine, or anticholin-ergics for a minimum of four weeks prior to inclusion.
* The following oral dopamine agonist drugs are allowed in this trial: pramipexol up to a total daily dose of 3,15mg, ropinirol up to a total daily dose of 24mg, cabergoline up to a total daily dose of 6mg or combinations Concomitant diseases are stable and well controlled Willingness and ability to comply with all trial requirements Written informed consent

Exclusion Criteria:

* Non-idiopathic Parkinson's disease (e.g. drug-induced or other forms of secondary or atypical parkinsonism such as MSA)
* Significant neurological symptoms not accounted for by Parkinson's disease
* History or presence of dementia demonstrated by the Mini-mental status examination (MMSE < 24)
* Presence of major depression according to DSM IV criteria (≥ 6 months)
* History or presence of epilepsy
* Presence of dopaminergic psychosis
* Unstable severe concomitant diseases (e.g. liver diseases, kidney diseases or clinically relevant cardiac or coronary dysfunction)
* Presence of heart valvular fibrosis or indication of significant valvular stenosis / insufficiency on echocardiogram
* History of syncope and/or severe or otherwise symptomatic orthostatic hypotension
* Present treatment with neuroleptics, including atypical neuroleptics
* Treatment with other CNS active drug therapy (e.g. sedatives, hypnotics, anti-depressants, anxiolytics) unless the dose has been stable for at least four weeks prior to the baseline visit
* Participation in another trial of an investigational drug within the last 28 days or current participation in another trial of an investigational drug
* Clinically significant laboratory abnormalities
* Previous neurosurgery for Parkinson's disease
* Alcohol or drug abuse in the past three years

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-07

PRIMARY OUTCOMES:
Change from baseline B0 to T6 in total daily "OFF-time and ON-time with troublesome dyskinesia

SECONDARY OUTCOMES:
Secondary objectives are to evaluate quality of life, quality of sleep, UPDRS Score
clinical global impression, safety and tolerability.
After the double-blind period, long-term efficacy of lisuride will be assessed for further 2 years in an open-label extension of the study

CONTACTS AND LOCATIONS:
Overall Officials: J. Winkler, Professor, Principal Investigator — Klinik und Poliklinik für Neurologie der Universität Regensburg
Locations (1):
- Imerem GmbH, Nuremberg, Germany